CLINICAL TRIAL: NCT02212366
Title: Enhancing Cognition in Patients With Late-Life Depression: A Randomized Controlled Trial of Transcranial Direct Current Stimulation
Brief Title: To Enhance Cognition in Late Life Depression Using Transcranial Direct Current Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Principal Investigator, Tarek Rajji, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 131/2013
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Cognition; Depression
Keywords: TDCS; Depression; Brain Stimulation; Memory; Cognition; EEG
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active TDCS (Experimental): 2-week course of daily (5 days/week) active bilateral anodal TDCS, duration 30 minute each session. Current 2 mA.
  Interventions: Device: Active TDCS
- Sham TDCS (Sham Comparator): 2-week course of daily (5 days/week) Sham bilateral tDCS. Duration 30 minute each session.
  Interventions: Device: Sham TDCS

INTERVENTIONS:
Device: Active TDCS — Active Stimulation
  Arms: Active TDCS
Device: Sham TDCS — Sham Stimulation
  Arms: Sham TDCS

SUMMARY:
Late Life Depression (LLD) is a serious health problem which not only causes depressed mood but also results in impairments in memory and attention. These impairments are likely to be resistant to treatment, which increases the chances of developing dementia even after successful treatment of mood.This study is a randomized controlled trial of transcranial Direct Current Stimulation (tDCS) in people with LLD to enhance their cognition after successful treatment of mood with established medications. tDCS is non invasive, relatively inexpensive and portable, and has been found to be safe.This study also serves as a pilot study to assess the effects of tDCS on cognition and neurophysiologic markers of cognition among patients with LLD. Primary study hypothesis is that participants Participants randomized to tDCS will perform better on a working memory task 2 weeks and 3 months following the tDCS course.

DETAILED DESCRIPTION:
tDCS is a non-invasive brain stimulation method that utilizes low intensity electrical current either to increase cortical excitability with an anodal electrode or to suppress cortical excitability with a cathodal electrode. tDCS produces its effects through long lasting changes in neuroplasticity: in animal studies, tDCS results in long-term potentiation and brain-derived neurotrophic factor secretion; in human studies, tDCS results in potentiation of neurophysiologic markers of neuroplasticity. Consistent with these preclinical findings, tDCS to the temporoparietal cortex or left DLPFC improves memory in patients with mild to moderate Alzheimer disease(AD). tDCS has also been tested among patients with depression - including by our group - but mainly as a treatment for depressive symptoms. In one recent large study one session of bilateral anodal tDCS was shown to enhance working memory among midlife participants with major depression prior to receiving any treatment. However, it is still not known (1) whether tDCS improves cognition beyond the partial improvement that is associated with resolution of depressive symptoms; or (2) whether it has a more fundamental and long lasting effect on cognition.

This trial will assess the acute and long-term effects of a 2-week course of daily (5 days/week) bilateral anodal tDCS of the DLPFC on cognition, and in particular working memory among 36 patients with LLD. We will recruit and randomize participants who have already been treated for LLD prior to consenting to the study and who still meet criteria for remission while on antidepressant medications.

This trial will also be used as a platform to explore the effect of tDCS on neurophysiologic measures of plasticity during working memory performance. Working memory is supported by re-entrant circuits, some are local within the DLPFC and others are long-range connecting the DLPFC to more posterior cortices. These networks result in high and low frequency neuronal oscillations that can be captured by electroencephalography (EEG). Using novel neurophysiologic analyses, our group and others have demonstrated that the modulation of high-frequency (particularly gamma) oscillations by low-frequency (particularly theta) oscillations - "theta-gamma coupling" - is a neurophysiologic marker of working memory. Thus, we will explore the effect of tDCS on theta-gamma coupling.

ELIGIBILITY:
Inclusion Criteria:

1. Women and men of any races or ethnicity
2. Age 60 and above
3. Major depressive disorder, single or recurrent per SCID DSM-IV criteria AND remission from that episode as defined by DSM IV-TR criteria for remission.
4. Montgomery-Asberg Depression Rating Scale (MADRS) score less than 10.
5. Ability to speak English fluently enough to complete all research assessments.
6. Corrected visual ability to read newspaper headlines; hearing capacity to respond to a raised conversational voice
7. Willingness and ability to provide consent

Exclusion Criteria:

1. DSM IV TR criteria for any dementia
2. DSM IV TR criteria for life-time bipolar disorder, schizophrenia, schizoaffective disorder, or other psychotic disorders
3. DSM IV TR criteria for any substance abuse or dependence within the past 6 months
4. Presence of psychotic features or any other symptoms that would make the participant unable to participate in the study.
5. Any medical contra-indications to tDCS.
6. Electroconvulsive therapy in the last 6 months.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-05; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
To compare performance on working memory task (N-Back) and neuropsychological battery between active and sham TDCS groups | Two weeks following the TDCS course

SECONDARY OUTCOMES:
To compare performance on working memory task (N-Back) and neuropsychological battery between active and sham TDCS groups | Three months following the TDCS course

OTHER OUTCOMES:
To compare theta-gamma coupling as measured by electroencephalography between active and sham TDCS groups. | Two weeks following the TDCS
To compare theta-gamma coupling as measured by electroencephalography between active and sham TDCS groups. | 3 months following the TDCS

CONTACTS AND LOCATIONS:
Overall Officials: Tarek K Rajji, MD, Principal Investigator — Center for Addiction and Mental Health
Locations (1):
- Center for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kumar S, Batist J, Ghazala Z, Zomorrodi RM, Brooks H, Goodman M, Blumberger DM, Daskalakis ZJ, Mulsant BH, Rajji TK. Effects of bilateral transcranial direct current stimulation on working memory and global cognition in older patients with remitted major depression: A pilot randomized clinical trial. Int J Geriatr Psychiatry. 2020 Oct;35(10):1233-1242. doi: 10.1002/gps.5361. Epub 2020 Jul 21. PMID 32525222